CLINICAL TRIAL: NCT00185718
Title: Impact of Treatment Induced Premature Menopause on Quality of Life Following Blood and Marrow Transplantation
Brief Title: Impact of Treatment Induced Premature Menopause on Quality of Life
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BMT160; 79700; BMT160; NCT00185718; 13644 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Menopause, Premature
MeSH Terms: conditions — Menopause, Premature

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To understand the impact of treatment induced menopause on quality of life and sexuality following blood and marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal
* sexually active women
* able to read and write English

Exclusion Criteria:

- postmenopausal females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women become menopausal as a result of BMT
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2003-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1 year
  To describe the impact of premature menopause on sexuality and quality of life.
Sexuality | 1 year
  To describe the impact of premature menopause on sexuality and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Karl G. Blume, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States